CLINICAL TRIAL: NCT05338606
Title: Expanded Access to Bimatoprost
Brief Title: Expanded Access to Bimatoprost (Durysta)
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C21-630
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Open-angle Glaucoma
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Bimatoprost Sustained Release Implant — Intraocular Implant
  Other Names: AGN-192024; Durysta

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to Durysta (Bimatoprost) prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* The participant must not be eligible for bimatoprost implant (Durysta) clinical trial.
* Eligibility for this program is limited to patients with moderate or worse glaucoma who are at risk of severe visual impairment based on physician assessment of risk factors associated with visual field progression as defined by the respective country/regional glaucoma clinical practice guidelines (eg, Canadian Ophthalmological Society guidelines, European Glaucoma Society guidelines, etc.), and who have exhausted all the appropriate pharmaceutical treatment options and are contraindicated for surgery, which may include:

  * Patients with ocular comorbidities such as severely scarred conjunctiva (eg, chemical burns, Stevens-Johnson Syndrome), scleral thinning.
  * Patients who are intolerant to any pre- , intra-, or post-op treatments (e.g allergy/intolerance to medical treatments or to anesthesia).
  * Patients with systemic comorbidities (e.g cardiovascular conditions) in which any surgery is not recommended

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie